CLINICAL TRIAL: NCT03673787
Title: Ice-CAP: A Phase I Trial of Ipatasertib in Combination With Atezolizumab in Patients With Advanced Solid Tumours With PI3K Pathway Hyperactivation
Brief Title: A Trial of Ipatasertib in Combination With Atezolizumab
Acronym: IceCAP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR4720
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor; Glioblastoma Multiforme; Prostate Cancer Metastatic
MeSH Terms: conditions — Glioblastoma | interventions — ipatasertib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I (Experimental): Increasing doses of ipatasertib in combination with a fixed dose of atezolizumab to establish the recommended phase II dose.
  Interventions: Drug: ipatasertib; Drug: Atezolizumab
- Phase II (Experimental): The Phase II part of the study will evaluate the recommended phase II dose of ipatasertib identified in Phase I, in combination with atezolizumab, in six patient cohorts: patients with solid tumours who have hyperactivation of the PI3K pathway; patients with castrate-resistant prostate cancer with PTEN loss; patients with glioblastoma; patients with melanoma; patients solid tumour types refractory to immune-checkpoint inhibitors; patients with gynaecological cancers.
  Interventions: Drug: ipatasertib; Drug: Atezolizumab

INTERVENTIONS:
Drug: ipatasertib — Ipatasertib will be supplied as film-coated tablets in two strengths (100 and 200 mg) differentiated by size, shape, and weight of tablets. Ipatasertib tablets are packaged in high-density polyethylene bottles with desiccant.
Drug: Atezolizumab — Atezolizumab will be supplied as a single-use 20 mL USP/Ph. Eur Type 1 glass vial as a colourless-to-slightly-yellow, sterile, preservative-free clear liquid solution intended for intravenous (IV) administration.

SUMMARY:
This is a single centre, proof-of-concept phase I trial of atezolizumab in combination with ipatasertib. There are two parts to this study, the dose escalation phase (Part A) and the dose expansion phase (Part B). Part A, will determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D). This will be followed by the Part B dose expansion phase to further characterise the safety and tolerability and to assess the pharmacodynamic activity of the combination.

DETAILED DESCRIPTION:
This is a Phase 1 trial of atezolizumab in combination with ipatasertib. There are two parts to this study. Part A: dose escalation, and Part B: dose expansion.

Part A:

The investigators will investigate the combination of a fixed dose of atezolizumab (1200mg) in combination with escalating doses of ipatasertib in patients with advanced solid tumours (Cohort A1) and patients with resectable glioblastoma multiforme (GBM) (Cohort A2).

Cohort A1 (advanced solid tumours):

There will be an ipatasertib run-in phase of 14 days of continuous oral dosing with paired pre and post-treatment blood and tissue samples. Combinations dosing will commence on Cycle 1 Day 1 with the atezolizumab infusion. Cycle 1 will therefore be 35 days. Only patients with advanced solid tumours recruited into Cohort A1 will be included in dose escalation decisions and determination of the MTD and recommended Phase 2 dose (RP2D) for part B.

Cohort A2 (potentially resectable GBMs):

There will be an ipatasertib run-in phase of at least 14 days and up to 21 days followed by surgical resection of the patient's tumour (5 day window for surgery). Ipatasertib dosing will be stopped 48 hours prior to surgery and combination dosing on Cycle1Day1 (C1D1) will commence after recovery. Accrual to Cohort A2 will run in parallel Cohort A1 without formal dose escalations and patients in Cohort A2 will not be included in dose escalation decisions for Cohort A1.

Recruitment to Part A is complete.

Part B:

Patients will be enrolled into the expansion phase (Part B) to further characterize the tolerability of the RP2D (established in Cohort A1) of the combination in specific subgroups of patients. Part B of the study will have a pre-screening component for patients with solid tumours (Cohorts B1 and B2) to allow for enrichment for these specific subgroups of patients.

Part B of the study will have three cohorts:

* Cohort B1: patients with solid tumours with hyperactivation of PI3K pathway as determined by pathogenic mutations identified by next generation sequencing (NGS) (eg known activating mutations in PIK3CA, AKT1, AKT2) or PTEN loss (assessed by immunohistochemistry (IHC) (n=12).
* Cohort B2: patients with castrate-resistant prostate cancer with PTEN loss as assessed by IHC (n=12)
* Cohort B3: patients with glioblastoma (n=12) of which at least three (n=3) patients will have potentially resectable recurrent glioblastomas. Recruitment to cohort B3 is complete.
* Cohort B4: patients with melanoma post progression on immune-checkpoint inhibitors (n=12)
* Cohort B5: patients with other tumour types refractory to immune checkpoint inhibitors (where immune checkpoint inhibitors are licensed, e.g. bladder cancer, head and neck SCC, NSCLC) (n=12)
* Cohort B6: patients with gynaecological cancers (including ovarian cancer, cervical cancer, endometrial cancer) (n=12)

Approximately 12 patients with solid tumours and 3 patients with glioblastoma will be entered into Part A of this trial and a further 72 patients will be enrolled into part B of the trial for an expected maximum of 87 patients on the study. If the MTD is reached in Part A with less than 15 patients enrolled, the investigators may enrol further patients at the R2PD in Part A to a maximum of 15 patients to include sufficient numbers of patients for the proof-of-concept translational studies. Additional subjects may be enrolled in a given cohort to ensure that the required number of evaluable subjects in each cohort is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. PART A1: Patients with histologically or cytologically confirmed malignant advanced solid tumours refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient;

   PART A2: Patients with advanced glioblastoma with potentially surgically resectable disease.

   PART B1: Patients with histologically or cytologically confirmed malignant advanced solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient, with somatic mutations or other aberrations predicted to result in a hyperactivated PI3K-AKT pathway (eg activating mutations in PIK3CA, AKT1, AKT2) or PTEN loss (assessed by immunohistochemistry (IHC) (n=12).

   PART B2: Patients with histologically or cytologically confirmed malignant castrate refractory prostate cancer, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient, with PTEN loss confirmed by immunohistochemistry H-score <30 as established in our local laboratory PART B3: Patients with relapsed histologically confirmed glioblastoma. At least 3 patients will need to have potentially surgically resectable disease.
2. Part A1: Evaluable disease as assessed by immune-modified RECIST 1.1 (solid tumours).

   Part A2: Evaluable disease as assessed by Response-assessment in Neuro-Oncology (RANO) criteria for glioblastoma patients. Part B1: Measurable disease as assessed by immune-modified RECIST Part B2: Measurable disease as assessed by immune-modified RECIST 1.1 OR evaluable disease as per Prostate Cancer Working Group 3 (PCWG 3) criteria Part B3: Measurable disease as assessed by RANO
3. All patients with advanced solid tumours must be willing and able to have fresh paired tissue biopsies for biomarker analysis. All patients with potentially resectable glioblastomas being considered for Part A2 and Part B3 must be willing and able to have surgical resection with fresh tissue samples provided for translational studies.
4. Life expectancy of at least 12 weeks.
5. World Health Organisation (WHO) performance status of 0-1
6. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week prior to the first dose of either Investigational Medicinal Product (IMP)

   Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

   Either:

   Creatinine OR IF Creatinine > 1.5 times ULN then Calculated creatinine clearance <1.5 times ULN

   ≥ 50 mL/min (uncorrected value)

   Coagulation INR < 1.5 APTT <1.5x ULN (except for potentially resectable glioblastoma patients enrolled onto the surgical resection arms where the APTT should be <1.2x ULN Triglycerides ≤ 300 mg/dL Cholesterol ≤ 300 mg/dL

   7.18 years or over

8.Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up 9.Female patients with reproductive potential must have a negative serum pregnancy test within 14 days prior to start of trial.

Exclusion Criteria:

* 1.Radiotherapy, endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and four weeks for investigational medicinal products) before treatment, except for hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with castrate resistant prostate cancer, which are permitted, and bisphosphonates or RANK ligand antagonists that are permitted for the management of bone metastases.

  2.Ongoing Grade 2 or greater toxicities from pre-existing conditions or from previous treatments. Exceptions to this are alopecia.

  3.Clinically significant abnormalities of glucose metabolism as defined by any of the following:

  ◦Diagnosis of diabetes mellitus types I or II (irrespective of management).

  ◦Glycosylated haemoglobin (HbA1C) ≥7.50% at screening
  * Fasting Plasma Glucose ≥ 8.3mmol/L (150 mg/dL) at screening. Fasting is defined as no caloric intake for at least 8 hours.

    4.Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) from time of consent, during the trial and for six months afterwards are considered eligible.

    5.Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

    6.For patients with solid tumours, known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:
  * Evaluable or measurable disease outside the CNS is present.
  * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the baseline disease assessment
  * Not requiring corticosteroids.

    7.Major surgery within four weeks of the first dose of study treatment. 8.History of malabsorption syndrome or other condition that would interfere with enteral absorption.

    9.At high medical risk because of non-malignant systemic disease including active uncontrolled infection.

    10.Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).

    11.Has a known history of clinically significant liver disease, including viral or other hepatitis or cirrhosis.

    12.Has an active autoimmune disease that has required systemic treatment in past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with a history of inflammatory bowel diseases such as Crohn's disease or ulcerative colitis will be excluded from the study. Patients with Sjogren's syndrome will not be excluded from the study. In addition patients that experienced a Grade 2 or higher immune-related AE's on treatment with immunotherapy will be excluded from the study. Patients with inactive autoimmune disease which has previously required systemic therapy, may be considered on a case-by-case basis after discussion with the sponsor.

    13.Has a known history of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.

    14.Has a known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.

    15.Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the chief Investigator. Stable use (i.e., no change in dose within 1 month prior to Day 1 of Cycle 1 of inhaled corticosteroids is allowed.

In the Part B dose expansion only, patients with castrate-resistant prostate cancer who have been on long-term steroids, will be allowed, provided the average total daily dose of steroids for the two weeks prior to commencement of trial is ≤10mg prednisolone/day. Again, in the Part B3 dose expansion only, patients with glioblastoma will be allowed to be enrolled if they had been on a stable dose of steroids ≤3mg Dexamethasone for at least 5 days prior to Day 1 of Cycle 1.

16.Has received a live vaccine within 30 days of planned start of study therapy. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.

17.Any of the following cardiac criteria:

* Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms (ECGs) within 5 minutes of each other.
* Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete left bundle branch block, third degree heart block. Controlled atrial fibrillation is allowed.
* Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association [NYHA Grade 2]

  18.Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.

  19.Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for three years or more and are deemed at negligible risk for recurrence, are eligible for the trial.

  20.Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of ipatasertib and atezolizumab. Participation in an observational trial would be acceptable.

  21.Patients with prior exposure to a PI3K or AKT inhibitors will be excluded from this study. Patients with prior exposure to mTOR inhibitors will be permitted to be enrolled on study. Patients with prior exposure to immunotherapy (either CTLA-4, PD-1/PD-L1 inhibitor/cellular therapy) will be excluded from the dose escalation Part A of the study, but will be permitted to enrol onto the Part B dose expansion as long as they did not experience any ≥Grade 2 immune-adverse event toxicity while on their prior immunotherapy.

  22.Is taking or requiring the continued use of any of the prohibited concomitant medications listed in 5.8 Concomitant medication and treatment.

  23.Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To identify a maximum tolerated dose in Phase I | 12 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
To determine the number and type of treatment-related adverse events of the two drug combination as assessed by CTCAE v4.0 | 24 months
  Frequency and severity of treatment-emergent adverse events graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

SECONDARY OUTCOMES:
Determination of changes in immune-cell population in blood and plasma, using Fluorescence-Activated Cell Sorting (FACS) | 24 months
  The investigators aim is to analyse the changes in immune-cell population and look at the host immune cell cytokine profile using FACS
To assess the tumour microenvironment by immunophenotyping | 24 months
  Immunophenotyping can determine the changes in the tumour microenvironment, by looking at changes in tumour-infiltrating lymphocytes, myeloid derived suppressor cells (MDSCs) and regulatory T cells

OTHER OUTCOMES:
Characterisation of the pharmacodynamic profile of exploratory biomarkers using RNA sequencing. | 24 months
  Immune transcriptome profile changes will be looked at using Whole transcriptome sequencing. Exploratory biomarkers will be determined as the trial progresses.
Evaluation of disease response by immune-modified RECIST criteria version 1.1 | 24 months
  To obtain a preliminary assessment of antitumour activity of combination of atezolizumab with ipatasertib in patients with tumours exhibiting hyperactivation of the PI3K pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MRCP, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided